CLINICAL TRIAL: NCT04063410
Title: A Single-Institution, Single-Arm, Self-Controlled Trial Evaluating Perforator Phase Contrast Angiography (pPCA) as the Primary Preoperative Imaging Technique in Post-Mastectomy Breast Reconstruction Using Abdominal-Based Free Flaps
Brief Title: Evaluation of Perforator Phase Contrast Angiography in Developing Surgery Plans for Patients With Breast Cancer Undergoing Breast Reconstruction With Free-Flap Methods After Mastectomy
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: We are closing this study as our clinical partners have all relocate from OSU and we could not find continued interest. However, we demonstrated the feasibility of this imaging approach on which we also filed a patent.
Sponsor: University of Cincinnati (Other)
Responsible Party: Principal Investigator, Michael V Knopp MD PhD, Principal Investigator, University of Cincinnati
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: OSU-18094; NCI-2018-03417 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2019-08-19; First posted 2019-08-21 (Actual); Last update posted 2024-01-18 (Actual); Status verified 2024-01

CONDITIONS: Mammoplasty Patient
MeSH Terms: interventions — Cerebral Angiography

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- Screening (pPCA) (Experimental): Patients undergo standard of care CTA and undergo pPCA MRI for up to 60 minutes before surgery.
  Interventions: Procedure: Angiography; Procedure: MRI-Based Angiogram; Other: Quality-of-Life Assessment

INTERVENTIONS:
Procedure: Angiography — Undergo standard of care CTA
Procedure: MRI-Based Angiogram — Undergo pPCA
  Other Names: Magnetic Resonance Angiogram; MRA
Other: Quality-of-Life Assessment — Ancillary studies
  Other Names: Quality of Life Assessment

SUMMARY:
This phase II trial studies how well an imaging technique called perforator phase contrast angiography (pPCA) works in developing surgery plans for patients with breast cancer undergoing breast reconstruction after breast removal (mastectomy) using abdominal-based free flap methods. Free flaps are units of tissue transferred from one area of the body to another with an intact blood supply. pPCA uses magnetic resonance imaging (MRI) to create images of blood vessels inside the body. Using pPCA may help doctors develop better surgical plans for patients with breast cancer undergoing post-mastectomy reconstruction surgery with free flap methods.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To assess the quality of surgical plans prepared under the guidance of the non-contrast, ionizing-radiation-free perforator phase contrast angiography (pPCA) against plans based upon the current gold standard, the X-ray-based, contrast-enhanced computed tomographic angiography (CTA).

SECONDARY OBJECTIVES:

I. To assess whether pPCA is more accurate than CTA for vessel size measurement.

II. To assess the impact of pPCA-based surgical planning on the clinical outcomes of abdominal-based free flap surgery.

III. To obtain and analyze cost/expenditure information for pPCA-guided abdominal-based free flap procedures.

OUTLINE:

Patients undergo standard of care CTA and undergo pPCA MRI for up to 60 minutes before surgery.

After surgery, patients will be followed up at 24 hours, 1 week, 3 months, 1 year and 2 years.

ELIGIBILITY:
Inclusion Criteria:

* Subject must weigh =< 350 lbs.
* Subject must be scheduled to receive uni- or bilateral breast reconstruction using one of the abdominal-based free flap techniques (deep inferior epigastric perforator [DIEP] flap, superficial inferior epigastric artery [SIEA] flap, or free-transverse rectus abdominis musculocutaneous [TRAM] flap) within the next 12 months.
* Subject must have received, or be scheduled to receive at least one preoperative CTA prior to the surgery.
* Subject must be able to lie in both prone and supine positions for at least 30 minutes.

Exclusion Criteria:

* Subjects who are determined to be incompatible for MRI based on local policy.
* Subjects with previous history of abdominal-based free flap surgery.
* Severe anxiety or claustrophobia that would prohibit the required study procedures from being conducted.
* Any serious and/or unstable pre-existing medical disorder, psychiatric disorder, or other conditions that could interfere with the subject?s safety, the informed consent procedure, or compliance to the study protocol, in the opinion of the investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2023-01-01 (Estimated); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Occurrence rate of surgical plan scenarios | Up to 2 years
  When all participating plastic surgeons reach a consensus decision on the final surgical plan after jointly reviewing the perforator phase contrast angiography (pPCA)-based and contrast-enhanced computed (CTA) based preliminary plans, one of four scenarios may occur: I. The pPCA-based and CTA-based plans are identical. Both are accepted as the final plan; II. There is substantial discrepancy between the two preliminary plans. The pPCA-based plan is eventually accepted as the final plan; III. There is substantial discrepancy between the two preliminary plans. The CTA-based plan is eventually accepted as the final plan; IV. There is substantial discrepancy between the two preliminary plans, but neither the pPCA-based plan nor the CTA-based plan is deemed acceptable. The final plan is proposed based upon comprehensive assessment of both image sets. The occurrence rate of scenario I-IV cases will be estimated with 95% confidence interval, respectively.
Acceptance rate for pPCA-based surgical plans | Up to 2 years
  The acceptance rate for pPCA-based plans will be evaluated using one-sided non-inferiority test of correlated proportions with non-inferiority margin of 15%. Perforator size measurements obtained with pPCA or CTA will be summarized separately, and be compared between pPCA and CTA using paired t-test.
Postoperative major complication rate | At 2 years
  Will be calculated and exact binomial 95% confidence interval will be provided. The calculated major complication rate will be compared with historical data. The association of complications with demographic and clinical characteristics (e.g., age, obesity, laterality and radiation) will be explored using two sample t-test or Wilcoxon test for continuous variables, and chi-square test or Fisher?s exact test for categorical variables. Logistic regression model will also be used to study the association between the complications and the pPCA/CTA-based plans, controlling those significant confounders.
Quality of life questionnaire (BREAST-Q) | Baseline up to 2 years
  Patient reported outcome for breast reconstruction questionnaire (BREAST-Q) score for satisfaction with breast will be summarized using descriptive statistics (mean and standard deviation) at baseline, 1 year postoperative, 2 years postoperative, as well as the change from baseline to postoperative. BREAST-Q score at 2 years will be compared with historical data.

CONTACTS AND LOCATIONS:
Overall Officials: Michael Knopp, MD, Principal Investigator — Ohio State University Comprehensive Cancer Center
Locations (1):
- Ohio State University Comprehensive Cancer Center, Columbus, Ohio, United States

REFERENCES:
- See also: The Jamesline — http://cancer.osu.edu